CLINICAL TRIAL: NCT04615897
Title: Effectiveness of New Technologies in the Balance, Gait and Cognitive Function in Healthy Elderly
Brief Title: Efficiency of New Technologies in the Aging Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Maria LuIsa Benitez Lugo, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MLugo - USeville
Record Dates: First submitted 2018-03-06; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Aging
Keywords: gait; attention; memory

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental aging (Experimental): The subjects received 16 sessions (Two per week) of exercise with new tecnology between two measurements of the variable.
  Interventions: Procedure: new tecnology intervention
- Control Aging (No Intervention): The subjects doesn´t received 16 sessions (Two per week) of exercise with new tecnology between two measurements of the variable.

INTERVENTIONS:
Procedure: new tecnology intervention — The intervention consists of 16 sessions, performed with a frequency of twice a week, the final evaluation was made within three days after the end of the last treatment session. It is used for the motor task, the "Fishing Under Zero" exercise, included within the "balance" modality and the so-called "Step Plus" located in the aerobic exercise folder. Each subject carried out the training taking into account the following methodology: 3 cycles of the "Fishing under zero" exercise, one cycle of the "Step Plus" exercise and 3 cycles of the "Fishing under zero" exercise, the approximate duration of the task being about 30 minutes.
  Arms: Experimental aging

SUMMARY:
This study tries to analyze the effectiveness of the application of the new technology in the maintenance of an active time. To do this, the investigators performed a laboratory test where they evaluated the physical and cognitive variables before and after the intervention and analyzed the improvement in the psychocognitive abilities in the experimental group and the use of physical and cognitive functions in the control group.

DETAILED DESCRIPTION:
The main objective of this study is the demonstration of the effectiveness of a motor task, making use of the Nintendo Wii video game console, in healthy elderly people, as well as demonstrating the interaction between the physical and cognitive aspects and the decline that in these functions causes the aging process. Methodology: A double blind, controlled and randomized clinical trial was developed on a total sample of 46 subjects, with a mean age of 72.59 years. For the collection of data, the following evaluation scales and computerized tests were passed (Cognitive Miniexamen, Depression Scale, Berg Scale, Tinetti Scale, Timed Up and Go test, Oddball Test and the Attention Network Test).

ELIGIBILITY:
Inclusion criteria:

* Be 60 years old or older.
* Have compensated the auditory or visual deficits that could suffer
* Absence of musculoskeletal problems that hinder functionality

Exclusion criteria:

* Presents cognitive impairment
* Obtain values in the Geriatric Depression Scale> 9.
* Presenten pathologies where the development of a motor task is counterproductive
* Sleep less than 6 hours a day

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Attention | At the start and the end of the study (65 days)
  This variable is obtained by performing two tests designed to quantify this cognitive function, using the E-prime computer program. Both tests are developed in the psychophysiology laboratory of the University of Seville. The first is to complete the "Test Oddball" and the second the "Attention Network Test-ELDERLY". Both tests measure the reaction times, in seconds and, the precision, in percentages. It involves two continuous quantitative measurements.
Memory | At the start and the end of the study (65 days)
  This variable is obtained from the score obtained in the scale called Miniexamen Cognitive (MEC), in which the subject must: respond to a series of questions that we perform related to the orientation, try to set a series of three words that the evaluator says to remember them later, develop a series of calculations, and work on a series of aspects related to language and its construction. At the end of the test, the subject obtains a score that determines the presence or absence of a cognitive problem. We consider it as a discrete quantitative variable.
Balance | At the start and the end of the study (65 days)
  This variable is studied using the Berg scale, which allows to quantify the balance of the subject in different positions, obtaining a global score that guides us on the general state of the balance function and guides us on a wheelchair dependence, the use of some technical help or total independence for the development of the march. We consider it as a discrete quantitative variable
Gait | At the start and the end of the study (65 days)
  This variable is configured by the application of the "Timed up and Go test" scale, which quantifies the time the subject takes to get up from a chair, walk 3 meters and return back to the starting position. We consider this variable as continuous quantitative
Global autonomy and risk of falls | At the start and the end of the study (65 days)
  This variable is analyzed through the application of the Tinetti Scale, which evaluates in a single instrument the function of balance and gait, as well as the risk of falls that elderly people present. In this sense, we can consider that it evaluates global autonomy. We consider this variable as discrete quantitative.

CONTACTS AND LOCATIONS:
Overall Officials: Benitez Lugo, PhD, Principal Investigator — University of Seville

IPD SHARING:
Plan to Share IPD: No